CLINICAL TRIAL: NCT02120183
Title: Investigating the Effects of a Psycho-educational Support Group Therapy on Cancer Caregivers' Burden and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NR13NMR139MP
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: The Effect of a Psycho-education Support Group Therapy
Keywords: Caregivers; Quality of life; Neoplasms; Psychotherapy, group; Family; Adaptation, psychological; Psycho-educational support group therapy; Cancer patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Psycho-educational support group therapy (Experimental): 4 week psycho-educational support group focusing on topics specific to psychosocial and emotional aspects of the cancer caregiving role
  Interventions: Behavioral: Psycho-educational support group therapy

INTERVENTIONS:
Behavioral: Psycho-educational support group therapy — Weekly sessions lasting 60 minutes. Topics addressed each week:
  Week 1: Coping with the diagnosis of loved one and dealing with uncertainty
  Week 2: Caring for the carer 1: Feeding your body (self-care, stress management, mindfulness concepts)
  Week 3: Caring for the carer 2: Feeding your mind (challenging negative thinking habits)
  Week 4: The emotions of caregiving (handling emotional reactivity)

SUMMARY:
This is a study to determine the effectiveness of a Group Therapy that provides psycho-education and support for caregivers of cancer patients. Caregivers must be between 21 and 64 years of age and be willing to attend a one-hour a week program for four weeks. The sessions will be in English, and a set of questionnaires (demographic data, some information about your family member with cancer, and scales: Caregiver Quality of Life-Cancer Scale (CQOLC), Perceived Stress Scale and the Hospital Anxiety Depression Scale (HADS)) will be completed at the start, at 4 weeks, at 8 weeks and at 12 weeks. Some participants placed on a wait-list to start the Group Therapy 4 weeks later will also complete the set of questionnaires at this point. A Feedback and Satisfaction Questionnaire will be completed at the end of the 4 week program. In addition, at the end of the 4 week program, some participants will go through a 15-minute interview.

DETAILED DESCRIPTION:
Participants Study participants are caregivers, recruited from the Medical Oncology Clinic (under NCIS) at NUH.

Intervention and Evaluation of the Psycho-educational Support Group Therapy This is a pre and post-intervention study with a control group design. The strength of this design is its experimental nature but without randomization, thereby avoiding the problems related to randomization. Instead, a wait-list is used as the control group.

Consecutive family caregivers who agree to participate will be placed in the first group (Group 1a) till a group size of ten is reached. The next ten will be put on a wait-list and form the control group (Group 1b), who will still be able to benefit from the program at a later time. In this manner subsequent treatment and control groups will be recruited.

The Intervention consists of weekly Psycho-educational Support Groups focusing on topics specific to psychosocial and emotional aspects of the cancer caregiving role. The Intervention is over a short duration of 4 weeks so as to appeal to caregivers and reduce the attrition rate. The proposed intervention is exploratory in nature but is hypothesized to be beneficial in helping to recognize and handle the difficult and often tumultuous journey of cancer caregiving. The planned Intervention was developed in discussions and consensus views using the Delphi method and adapted the brief integrative psychological therapy developed by Kua et al and psycho-educational programs at overseas centres. The CQOLC, the Perceived Stress Scale, and the HADS will be administered to participants at 4 time points: T1 (week 0), T2 (end of week 4), T3 (end of week 8) and T4 (end of week 12). The fourth time point is to evaluate whether the effects of the intervention are sustained. A Satisfaction and Feedback Questionnaire will be administered to participants at T2, immediately upon completion of the intervention. Some participants who have gone through the program will be invited to take part in a 15 minute interview. The purpose of the interview is to obtain feedback on the ways in which the program has been beneficial. The participants in the control group will complete a set of the same questionnaires when they are entered into the wait list; they will complete the questionnaires 5 times.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 64 years of age
* Willingness to attend a 1-hour program every week for 4 weeks
* Able to understand and speak basic English
* Able to understand and complete self-report questionnaires with minimal assistance
* Be the primary adult family member who provides care and support for the patient and lives together with the patient

Exclusion Criteria:

* Younger than 21 years of age, or 65 years of age and older
* Unable to understand and speak basic English
* Unable to understand and complete self-report questionnaires with minimal assistance

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Caregiver Quality of Life Index - Cancer | 4 weeks
Perceived Stress Scale | 4 weeks
Hospital Anxiety and Depression Scale | 4 weeks
Basic Psychological Needs Scale | 4 weeks
Healthcare Climate Questionnaire | 4 weeks
Perceived Competence Scale | 4 weeks
Interpersonal Support Evaluation List | 4 weeks
Benefit Finding | 4 weeks
Satisfaction and Feedback Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, Principal Investigator — Department of Psychological Medicine, National University Health System
Locations (1):
- National University Cancer Institute, Singapore, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Stenberg U, Ruland CM, Miaskowski C. Review of the literature on the effects of caring for a patient with cancer. Psychooncology. 2010 Oct;19(10):1013-25. doi: 10.1002/pon.1670. PMID 20014159
- [Background] Soothill K, Morris SM, Harman JC, Francis B, Thomas C, McIllmurray MB. Informal carers of cancer patients: what are their unmet psychosocial needs? Health Soc Care Community. 2001 Nov;9(6):464-75. doi: 10.1046/j.0966-0410.2001.00326.x. PMID 11846826
- [Derived] Mahendran R, Lim HA, Tan JY, Ng HY, Chua J, Lim SE, Kua EH, Griva K. Evaluation of a brief pilot psychoeducational support group intervention for family caregivers of cancer patients: a quasi-experimental mixed-methods study. Health Qual Life Outcomes. 2017 Jan 23;15(1):17. doi: 10.1186/s12955-017-0595-y. PMID 28114962
- [Derived] Mahendran R, Tan JY, Griva K, Lim HA, Ng HY, Chua J, Lim SE, Kua EH. A pilot, quasi-experimental, mixed methods investigation into the efficacy of a group psychotherapy intervention for caregivers of outpatients with cancer: the COPE study protocol. BMJ Open. 2015 Nov 19;5(11):e008527. doi: 10.1136/bmjopen-2015-008527. PMID 26586322